CLINICAL TRIAL: NCT02275793
Title: The Regulation of Pulmonary Vascular Resistance in Patients With Heart Failure
Acronym: PVR
Status: Completed | Type: Observational
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Other Study IDs: PVR
Record Dates: First submitted 2013-12-11; First posted 2014-10-27 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Diastolic Heart Failure; Pulmonary Hypertension
MeSH Terms: conditions — Heart Failure, Diastolic; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA storage for future exploratory research into genes/genetic variations which may indicate the presence or absence of pulmonary hypertension and congestive heart failure either as an extension of this research protocol or future protocols developed in the study of pulmonary hypertension/chf
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- high PH and normal PVR: Group I, diastolic heart failure with high PH and normal PVR
- high PH and high PVR: Group II, diastolic heart failure with high PH and High PVR
- normal PH and normal PVR: Group III, no heart failure, normal PH and normal PVR

SUMMARY:
Peripheral blood and blood following a pulmonary wedge pressure will be obtained from patients undergoing right heart catheterizations.

DETAILED DESCRIPTION:
It is well known that left sided heart disease can lead to pulmonary hypertension via a number of proposed mechanisms. The purpose in this study is to identify biomarkers in pulmonary hypertension to further understand the pathophysiology of this disease in patients with heart disease.Patients are recruited in the cardiac catheterization lab, which are undergoing right heart catheterization as per their plan of care established by their primary cardiologist. During the procedure, we will ask the performing cardiologist to obtain a blood sample of 40-50 milliliters from the catheter that they are using during the procedure. These blood samples will be sent for analysis of biomarkers. The patient will then have an echocardiogram done 1 year from their heart catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Ability to provide informed consent.
* Presenting for cardiac catheterization for evaluation of heart disease
* Ejection Fraction > 50%

Exclusion Criteria:

* Unable to provide informed consent.
* Unable or unwilling to comply with the protocol and follow up.
* Infiltrative cardiomyopathy
* Constrictive pericarditis
* Severe valvular disease
* Comorbid status with life expectancy <3 years
* Right ventricular dysplasia
* Congenital heart disease
* On immunosuppressive drugs.
* Patients who has heart transplant.
* Ejection Fraction < 50%
* Mean Pulmonary Artery Pressure <25
* Wedge pressure <15

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will study a cohort of patients that will be recruited from the cath lab during diagnositic heart catheterization
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-09; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 year
  Checking vital statistics on each patient at one year

SECONDARY OUTCOMES:
Morbidity | 1 year
  Checking vital statistics on each patient at one year

CONTACTS AND LOCATIONS:
Overall Officials: Samer Khouri, MD, Principal Investigator — University of Toledo Health Science Campus
Locations (1):
- University of Toledo, Health Science Campus, Toledo, Ohio, United States